CLINICAL TRIAL: NCT02430857
Title: Osteopathy and Latent Hypothyroidism: Effectiveness of Osteopathic Treatment on TSH in Patients With Latent Hypothyroidism
Brief Title: Osteopathy and Latent Hypothyroidism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Emanuel Amier Diekmann (Individual)
Responsible Party: Sponsor-Investigator, Emanuel Amier Diekmann, DO, Diekmann, Emanuel Amier
Organization: Diekmann, Emanuel Amier (Individual)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-5-2015
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Latent Hypothyroidism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OMT-Group (Experimental): The OMT-group will get an osteopathic treatment once a week for 1 hour for 5 weeks. The blood will be screened again after the treatment.
  Interventions: Other: OMT
- Controll Group (No Intervention): This group will receive no treatment. A blood screening is made again after 5 weeks.

INTERVENTIONS:
Other: OMT — Manuel osteopathic treatment of the spine
  Arms: OMT-Group

SUMMARY:
This study evaluates the effectiveness of stimulating the neurological segments c8-th5 in patients with latent hypothyroidism.

One half of the participants will receive an osteopathic manuel treatment in order to stimulate the relevant segments, the other half will receive no treatment.

DETAILED DESCRIPTION:
Patients with latent hypothyroidism show an increased hormone status in TSH and a normal hormone status in fT4. A study has shown that osteopathic treatment had positive effects to some symptoms in patients with latent hypothyroidism. The study was using the pain inventory as the instrument to measure the effect. In this study we want to evaluate the effectiveness of the treatment on the hormone status (TSH, fT4) The intervention group will receive a neurological osteopathic stimulation over 5 weeks. A parallel control group will not receive any therapy.

A follow up blood screening (TSH, fT4) will be done. The results of both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* latent hypothyroidism

Exclusion Criteria:

* Factors that Alter Thyroxine and Triiodothyronine Binding in Serum
* Increased thyroxin-binding globulin
* Decreased thyroxin-binding globulin
* Binding inhibitors
* Inherited Salicylates
* Pregnancy
* Androgens
* Furosemide
* Neonatal state
* Anabolic steroids
* Free fatty acids
* Estrogens
* Glucocorticoids
* Phenytoin
* Hepatitis
* Severe illness
* Carbamazepine
* Porphyria
* Hepatic failure
* nonsteroidal antiinflammatory drug (variable, transient)
* Heroin
* Nephrosis
* Heparin
* Methadone
* Nicotinic acid
* Mitotane L-Asparaginase
* 5-Fluorouracil
* SERMS (e.g., tamoxifen, raloxifene)
* Perphenazine
* spinal pathologies

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in TSH Concentration | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Diekmann, DO, Principal Investigator — Praxis fuer Osteopathy